CLINICAL TRIAL: NCT00378937
Title: An Open, Randomized, Parallel Group Study in Patients With Cancer Pain, To Compare a Two-Step Analgesic Ladder (Non-Opioid to Oxycodone) With Conventional Management Using A Three-Step Approach
Brief Title: Oxycodone or Standard Pain Therapy in Treating Patients With Cancer Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CRUK-ON/2003/1772; CDR0000507650 (Registry Identifier: PDQ (Physician Data Query)); EU-20640; EUDRACT-2004-004235-66; NAPP-CRUK-ON/2003/1772
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2007-07

CONDITIONS: Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Codeine; Levopropoxyphene; Morphine; Oxycodone

INTERVENTIONS:
Drug: acetaminophen
Drug: codeine phosphate
Drug: dextropropoxyphene hydrochloride
Drug: morphine sulfate
Drug: oxycodone hydrochloride
Procedure: management of therapy complications
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Oxycodone helps lessen pain caused by cancer and may improve quality of life. It is not yet known whether oxycodone works better and is more cost effective than standard therapy in treating patients with cancer pain.

PURPOSE: This randomized phase IV trial is studying oxycodone to see how well it works compared with standard pain therapy in treating patients with cancer pain and if it is more cost effective than standard pain therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall pain management in patients with cancer-related pain treated with oxycodone hydrochloride vs standard three-step analgesic therapy.
* Compare the health economics of these regimens in these patients.

Secondary

* Explore the factors that inform patients' decisions about commencing opioid analgesia.

OUTLINE: This is an open-label, multicenter, randomized, parallel group, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive an analgesic regimen, according to their level of pain, for up to 18 weeks.

  * Step 1: Patients in mild pain receive oral acetaminophen 4 times daily.
  * Step 2: Patients in mild-to-moderate pain receive oral codeine or oral dextropropoxyphene hydrochloride 4 times daily and oral acetaminophen 4 times daily.
  * Step 3: Patients in moderate-to-severe pain receive oral morphine or oral oxycodone hydrochloride 6 times daily (every 4 hours) with or without a non-opioid analgesic.

Patients may also receive an adjuvant drug (i.e., for side effects or for primary indication other than pain management that is analgesic in selected circumstances).

* Arm II: Patients receive oral oxycodone hydrochloride twice daily for up to 18 weeks. Patients may receive a different opioid analgesic or analgesia or adjuvant medication as in arm I, if needed.

Patients in both arms may also receive additional medication for breakthrough pain.

Patients complete a patient-assessment booklet (PAB) daily which includes a Box-Scale (BS)-11 rating for average pain; questions regarding contact (e.g., telephone or visit) with healthcare professionals on that day; and information regarding the number of times escape medication is used.

Quality of life and levels of cancer pain are assessed using the short form of the Brief Pain Inventory (BPI).

After completion of study treatment, patients are followed at 4 weeks.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Requires regular step-2 analgesia for the management of cancer-related pain

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Must be able to take oral medication
* Must be willing and able to complete a daily patient assessment booklet (PAB)
* No history of the following conditions:

  * Depression
  * Personality disorders that may lead to self-harm
  * Admission to the hospital for psychiatric reasons
  * Any other psychological disorder that, in the opinion of the investigator, would preclude study treatment
* Not at risk of additional CNS depressant effects due to study drugs
* No known history of alcohol or drug abuse or, in the opinion of the investigator, tendency towards drug abuse or addiction
* No current abuse of alcohol or drugs
* No known sensitivity to oxycodone hydrochloride or other opioids
* No history of a specific or allergic reaction to study drugs
* No contraindications as a result of adverse drug reaction or drug interactions of oxycodone or other opioid drugs
* No other condition that, in the opinion of the investigator, would make the patient unsuitable for study participation

PRIOR CONCURRENT THERAPY:

* More than 30 days since prior and no concurrent chemotherapy or radiotherapy
* At least 2 weeks since prior regular (i.e., 4 times per day) step-2 analgesics
* More than 3 months since prior regular use of opioids, defined as having a regular prescription of an opioid medication
* Not planning to undergo cancer-related surgery
* No other concurrent opioid-based medication other than oxycodone hydrochloride capsules as escape medication (arm II)
* No concurrent participation in another clinical trial involving a new chemical entity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-01; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Percentage of time in assessment periods 1 and 2 (i.e., first 4 weeks) with a Box-Scale (BS)-11 pain score of ≤ 4 (i.e., mild pain)

SECONDARY OUTCOMES:
Percentage of time in assessment periods 3 and 4 with a BS-11 pain score of ≤ 4
Mean BS-11 pain scores
Time to reach stable pain control
Mean escape medication use
Quality of sleep
Global assessment of pain relief with study drugs
Mean pain intensity, pain interference, and pain relief scores as measured by the Brief Pain Inventory
Overall number of phone calls, home visits by a nurse, home visits by a doctor, and unscheduled visits to a healthcare provider, related to pain control or analgesic medication during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Hanks, MD, Study Chair — University Hospitals Bristol and Weston NHS Foundation Trust